CLINICAL TRIAL: NCT05049551
Title: Quantitative Analysis of 99mTc-Pertechnetate Thyroid Uptake With a Large Field CZT Gamma Camera: Feasibility and Comparison Between SPECT/CT and Planar Acquisitions
Brief Title: Thyroid Uptake Quantification on a New Generation of Gamma Camera
Acronym: QUANTHYC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: 21-09
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Hyperthyroidism
Keywords: thyroid; uptake; quantification; CZT; Planar; SPECT/CT
MeSH Terms: conditions — Hyperthyroidism; Thyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to evaluate the potential of a new large field CZT gamma camera to estimate the thyroid uptake (TU) on Single photon emission computed tomography (SPECT) and SPECT/CT images in comparison with standard planar scintigraphy.

The secondary objective is to analyze the diagnostic contribution of SPECT/CT imaging.

DETAILED DESCRIPTION:
Planar and SPECT/CT scintigraphy will be performed on a new generation large field CZT gamma camera and thyroid uptake (TU) value will be calculated on planar acquisition for 23 consecutive patients referred in our department for hyperthyroidism.

With a quantitative approach using attenuation, scatter correction and iterative algorithm with resolution recovery we will have the possibility to calculate the TU value with SPECT or SPECT/CT acquisitions.

Our primary objective will be to evaluate the potential of a new large field CZT gamma camera to estimate the thyroid uptake on SPECT (Tomography without attenuation correction) and SPECT/CT (tomography with attenuation correction) acquisitions compared with standard planar scintigraphy as a gold standard.

The secondary objective will be to analyze the diagnostic contribution of SPECT/CT images.

To established this study it will be necessary to introduce cross-calibration factors performed from a thyroid phantom, for planar and SPECT acquisitions, to estimate the thyroid uptake values.

ELIGIBILITY:
Inclusion Criteria:

* Hyperthyroidism confirmed by blood test (TSH) and thyroid ultrasound

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-three consecutive participants referred in our nuclear medicine department for hyperthyroidism
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Thyroid uptake | Inclusion
  Quantification of thyroid uptake

SECONDARY OUTCOMES:
SPECT/CT | Inclusion
  Diagnostic contribution of SPECT/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ritt P, Vija H, Hornegger J, Kuwert T. Absolute quantification in SPECT. Eur J Nucl Med Mol Imaging. 2011 May;38 Suppl 1:S69-77. doi: 10.1007/s00259-011-1770-8. Epub 2011 Apr 12. PMID 21484383
- [Background] Gnesin S, Leite Ferreira P, Malterre J, Laub P, Prior JO, Verdun FR. Phantom Validation of Tc-99m Absolute Quantification in a SPECT/CT Commercial Device. Comput Math Methods Med. 2016;2016:4360371. doi: 10.1155/2016/4360371. Epub 2016 Dec 14. PMID 28096891
- [Background] Giovanella L, Avram AM, Iakovou I, Kwak J, Lawson SA, Lulaj E, Luster M, Piccardo A, Schmidt M, Tulchinsky M, Verburg FA, Wolin E. EANM practice guideline/SNMMI procedure standard for RAIU and thyroid scintigraphy. Eur J Nucl Med Mol Imaging. 2019 Nov;46(12):2514-2525. doi: 10.1007/s00259-019-04472-8. Epub 2019 Aug 7. PMID 31392371
- [Background] Mariani G, Tonacchera M, Grosso M, Orsolini F, Vitti P, Strauss HW. The Role of Nuclear Medicine in the Clinical Management of Benign Thyroid Disorders, Part 1: Hyperthyroidism. J Nucl Med. 2021 Mar;62(3):304-312. doi: 10.2967/jnumed.120.243170. Epub 2020 Oct 2. PMID 33008929
- [Derived] Serrano B, Amblard R, Beaumont T, Hugonnet F, Dietz M, Berthier F, Garnier N, Villeneuve R, Nataf V, Mocquot F, Montemagno C, Faraggi M, Paulmier B. Quantitative analysis of 99mTc-pertechnetate thyroid uptake with a large-field CZT gamma camera: feasibility and comparison between SPECT/CT and planar acquisitions. EJNMMI Phys. 2023 Jul 31;10(1):45. doi: 10.1186/s40658-023-00566-3. PMID 37522931